CLINICAL TRIAL: NCT03610373
Title: Personalizing Treatment Through Shared Decision Making for Youth Psychotherapy
Brief Title: Testing Psychosocial Treatment Planning Methods for Youth Anxiety and Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, David A. Langer, Research Associate Professor, Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 3462; K23MH101238 (NIH)
Record Dates: First submitted 2018-06-29; First posted 2018-08-01 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Anxiety Disorders; Depressive Disorder
Keywords: anxiety; depression; childhood; therapy; treatment; medical decision making
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder; Depression

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to receive a treatment planned primarily by the clinician (clinician guided) or planned collaboratively by the clinician, parent, and child (shared decision-making).
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessors do not have access to data regarding which arm each participant is in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shared Decision Making (Experimental): In this arm, parents and children will participate in a shared decision-making protocol with the clinician to plan their treatment. The treatment options available are established, evidence-based treatment techniques. The shared decision-making protocol was developed for this research project.
  Interventions: Behavioral: Modular Approach to Therapy for Children (MATCH)
- Clinician Guided (Active Comparator): In this arm, the clinician will plan the treatment in consultation with their supervisor, and share the treatment plan with the parent and child. The parent and child will have the opportunity to ask questions about the treatment plan (and, if they do not agree, reject the treatment plan), but they are not actively involved in making each decision. This is more typical of usual care.
  Interventions: Behavioral: Modular Approach to Therapy for Children (MATCH)

INTERVENTIONS:
Behavioral: Modular Approach to Therapy for Children (MATCH) — MATCH is a collection of 31 modules that correspond to the treatment procedures included in standard evidence-based treatments for youth depression, anxiety, and behavioral disorders.

SUMMARY:
Youth depression and anxiety represent a serious public health concern, with affected youth often experiencing social, familial, and academic impairment. Research evidence supports a growing array of effective treatments for youth depression and anxiety, yet as the collection of evidence-based treatments expands, so do the challenges of utilizing the evidence: clinicians must be able to (1) access, integrate, and apply the available evidence, and (2) engage in a collaborative process with each family to develop a plan that is responsive to each family's unique characteristics, preferences, and goals. Engaging caregivers and youths as active collaborators in the treatment planning process is a patient-centered approach with the potential to improve the process and outcome of youth mental health care by facilitating the personalization of established evidence-based treatment approaches. Such collaboration, frequently referred to as shared decision-making (SDM), is a hallmark of evidence-based practice and a key feature of federal guidelines for health care delivery. However, despite growing rhetorical support for SDM, empirical support is lacking, particularly in the area of youth mental health treatment. The absence of such research is unfortunate, given the potential for SDM to facilitate the dissemination and implementation of evidence-based treatments, and to personalize the use of established treatments to increase acceptability, retention, satisfaction, and overall effectiveness.

The present project tests the feasibility and acceptability of SDM through a pilot randomized controlled trial of 40 youths (ages 7-15) meeting diagnostic criteria for an anxiety or depressive disorder. The trial will compare an evidence-based treatment that is planned collaboratively with youths and caregivers using the SDM protocol, to an evidence-based treatment that is planned by the clinician and supervisor using pretreatment assessment data. Eligible youths will received up to 26 treatment sessions at no cost and complete assessments prior to the start of treatment, at the end of treatment, and six months following the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* a current DSM-5 principal diagnosis of a Major Depressive Disorder, Dysthymic Disorder, Generalized Anxiety Disorder, Separation Anxiety Disorder, Social Phobia, or Specific Phobia
* if receiving psychiatric medication, dose will be stable for at least 3 months at enrollment with ability to maintain medication
* youth and caregiver speak fluent English

Exclusion Criteria:

* active suicidality
* history of severe physical or mental impairments (e.g., mental retardation, autism spectrum disorders) in youth or caregiver
* participation in additional psychosocial treatment

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2016-10-04 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2019-08-27 (Actual)

PRIMARY OUTCOMES:
Anxiety Disorders Interview Schedule for DSM-IV - Child/Parent | Through completion of treatment, anticipated to be an average of 5 months
  The Anxiety Disorders Interview Schedule for DSM-IV - Child/Parent is an extensively tested semi-structured interview assessing the major anxiety, mood, and externalizing disorders.

SECONDARY OUTCOMES:
Satisfaction with Decision Scale | At the start of treatment, anticipated to be an average of 3 weeks after the initial assessment
  The 6-item Satisfaction with Decision Scale assesses satisfaction with treatment-related decisions. The scale score ranges from 6 (very low satisfaction) to 30 (very high satisfaction).

CONTACTS AND LOCATIONS:
Overall Officials: David A Langer, Ph.D., Principal Investigator — Boston University
Locations (1):
- Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided